CLINICAL TRIAL: NCT03990870
Title: Wiring Adolescents With Social Anxiety Via Behavioral Interventions (WASABI): a Closed-loop Mobile Intervention to Reduce Social Anxiety and Improve Social Skills
Brief Title: Wiring Adolescents With Social Anxiety Via Behavioral Interventions
Acronym: WASABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Minnesota (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSC-1016-19; 1R43MH121209-01 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Social Anxiety

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): dCBGT + WASABI
  Interventions: Other: dCBGT + WASABI
- Active Comparator (Active Comparator): dCBGT Only
  Interventions: Other: dCBGT Only

INTERVENTIONS:
Other: dCBGT + WASABI — Participants in the experimental treatment group will complete daily Ecological Momentary Assessments (EMAs), 1 hour of digitally delivered Cognitive Behavioral Group Therapy (dCBGT) per week, and weekly cognitive biases assessments and self-reports for 16 weeks. Participants assigned to this intervention will also have daily access to 1:1 and group chat Instant Messaging (IM) and will have weekly electronic check-ins with study staff (as needed).
  Arms: Experimental Treatment
Other: dCBGT Only — Participants in the active comparator group will be asked to attend 1 hour of digitally delivered Cognitive Behavioral Group Therapy (dCBGT) per week for 16 weeks and weekly electronic check-ins with study staff (as needed).
  Arms: Active Comparator

SUMMARY:
This study is a validation study to evaluate the acceptability, feasibility and impact of WASABI (Wiring Adolescents With Social Anxiety via Behavioral Interventions), a mobile application employing a closed-loop technology in adolescents with a Social Anxiety and to prepare for a large-scale efficacy trial in this population. The goal of this study is to evaluate WASABI-a clinician-assisted, adjunct to treatment, mobile application designed to augment the efficacy of psychological Evidence Based Treatments through a closed-loop technology.

DETAILED DESCRIPTION:
This study will employ an innovative and evidence-based mobile intervention that includes Ecological Momentary Assessments (EMAs) data collected from mobile devices, the WASABI closed-loop algorithm to detect exacerbation of social anxiety, and 1:1 and group-based videoconferencing and Instant Messaging with peers and providers. This study will test WASABI as an adjunct to digital Cognitive Behavioral Group Therapy (dCBGT) in adolescents with Social Anxiety (SA), in a parallel arm, double-blind, randomized, controlled clinical trial to assess feasibility and initial efficacy, to investigate the generalization of trained cognitive skills in the natural environment and improving anxiety and social functioning, and to prepare for a large-scale efficacy trials in adults with adolescents with Social Anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Potential participant is between the ages of 14 and 18 (inclusive) at the time of consent
2. Potential participant has a clinical diagnosis of Anxiety Disorder, as confirmed using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID), a brief structured diagnostic interview using Diagnostic and Statistical Manual of Mental Disorders-4 (DSM-IV) criteria
3. Potential participant has clinically significant Social Anxiety, as defined by a score of 25 or greater on the Social Phobia and Anxiety Inventory
4. Potential participant is clinically stable at time of screening as determined by the screening clinician/study team and the following criteria:

   * Potential participant has not experienced a psychiatric hospitalization within the 4 weeks prior to screening
   * Potential participant on a medication for anxiety and psychiatric disorders must be on a stable medication regimen for ≥ 4 weeks prior to screening, based on self-report.
5. Potential participant has a IQ Score > 80 as determined by performance on the Wechsler Abbreviated Scale of Intelligence (WASI-II)
6. Potential participant is a fluent English speaker, based on participant and/or parent/legal guardian self-report and as determined by the screening clinician, to ensure reasonable neuropsychological results on key assessments
7. Potential participant has adequate sensorimotor capacity to perform the intervention and study activities, including visual capacity adequate to read from a computer screen or mobile device at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control and use a mobile device and/or computer, based on participant and/or parent/legal guardian self-report and as determined by the screening clinician and/or study team
8. Potential participant has reliable access to wireless Internet connectivity
9. Potential participant can use iOS mobile applications

Exclusion Criteria:

1. Potential participant has a diagnosis of autism spectrum disorders, history of seizure disorder or seizure episodes within the last 2 years
2. Potential participant is currently receiving psychotherapy
3. Potential participant has a history of mental retardation, pervasive developmental disorder, head trauma, traumatic brain injury, or other neurological disorder that impairs cognition
4. Potential participant has medical illnesses deemed to interfere with participation in study activities and/or unstable and/or untreated conditions that may affect cognition, including substance abuse/dependence disorders, cardiovascular, endocrine, ongoing chemotherapy or other cancer treatment
5. Potential participant has history or current DSM-5 diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, delusion disorder, psychotic disorder NOS (not otherwise specified), bipolar disorder, substance dependence (<1 year), and/or mood congruent or mood incongruent psychotic features or disorders
6. Potential participants had significant medication changes, including changes to anxiety medications or other psychiatric medications, in the 4 weeks prior to screening
7. Potential participants who have answered 'yes' to:

   1. Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS), or,
   2. Any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the C-SSRS "Suicidal Behavior" portion will be excluded from the study if the ideation or behavior occurred within 2 months from Participant's date of consent (as recommended by the FDA for treatment trials.) Participants excluded for this reason will be referred for appropriate treatment. Further, the C-SSRS form will also be administered to all participants at the follow-up visit. Participants meeting these criteria at any time throughout the study will be asked to complete a final assessment, if appropriate, then withdrawn from the study and referred for appropriate treatment.
8. Potential participant that shows signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit or dCBGT session. Such participants will have that visit re-scheduled; participants with this problem occurring more than once may be excluded and dropped at the discretion of the PI.
9. Potential participant has problems performing assessments or comprehending or following spoken instructions, or participant displays behaviors during assessments visits or dCBGT sessions that, in the judgment of the clinician and study team, are likely to present significant problems for the Site Study personnel or other participants.
10. Potential participant is enrolled in a concurrent clinical trial involving an investigational pharmaceutical, medical device, behavioral treatment, or any other clinical trial that could affect the outcome of this study. However, participation in standard treatments (e.g., occupational therapy) or use of prescribed medications is allowable.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Biagianti, MD, Principal Investigator — Posit Science Corporation
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 participants were consented for this trial. Of those, 9 participants did not meet the inclusion criteria and one participant was no longer interested in participating in the study, prior to group assignment.
Period: Overall Study
Arm/Group | Experimental Treatment | Active Comparator
Started | 16 | 8
Completed | 13 | 7
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Treatment | Active Comparator | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 6 | 18
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.56 (1.63) | 16.38 (1.60) | 15.83 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 7 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Highest Grade Level Completed [Mean (Standard Deviation); unit: grade level] — This is the highest grade level completed in school.
  grade level | 9.13 (1.63) | 9.88 (1.89) | 9.38 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Ecological Momentary Assessment (EMA) Adherence
Description: Completed Ecological Momentary Assessments (EMAs) at least once per week. EMAs are repeated measures of the participants' current behaviors and experiences in real time.
Time Frame: 16 weeks
Population: Data was only collected from the dCBGT+WASABI group (Experimental Treatment group).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 13
percentage of participants | 53

2. Primary Outcome: Number of Group Sessions Attended
Description: Engagement with dCBGT (digitally delivered Cognitive Behavioral Group Therapy) and IM (Instant Messaging) will be evaluated.
Time Frame: 16 weeks
Population: While instant messaging was available to all study participants, no use was reported.
Measure: Mean (Standard Error); unit: group sessions attended
Arm/Group | Experimental Treatment | Active Comparator
Number analyzed (Participants) | 13 | 7
group sessions attended | 11.2 (1.0) | 10.7 (1.3)
Statistical Analysis 1: Comparison: Experimental Treatment vs Active Comparator; Test type: Superiority; p = 0.58, t-test, 2 sided

3. Primary Outcome: Ecological Momentary Assessments (EMA) Completion Rate
Description: The completion rate for Ecological Momentary Assessments will be evaluated. EMAs are repeated measures of the participants' current behaviors and experiences in real time.
Time Frame: 16 weeks
Population: Data was only collected from the dCBGT+WASABI group (Experimental Treatment group).
Measure: Median (Inter-Quartile Range); unit: number of entries
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 13
number of entries
  EMA Positive Thoughts | 12 [5 to 24]
  EMA Negative Thoughts | 10 [5 to 18.5]
  EMA Positive Feelings | 14 [4.5 to 24]
  EMA Negative Feelings | 14 [4.5 to 24]
  EMA Goals | 13 [4.5 to 23]

4. Primary Outcome: Percentage of Participants Who Completed the Social Phobia and Anxiety Inventory - Brief
Description: The completion rate for the Social Phobia and Anxiety Inventory - Brief will be evaluated.
Time Frame: 16 weeks
Population: Data was only collected from the dCBGT+WASABI group (Experimental Treatment group).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 13
percentage of participants | 69

5. Primary Outcome: Total Number of Participants Who Complete the Intervention
Description: The program completion rate will be evaluated.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment | Active Comparator
Number analyzed (Participants) | 16 | 8
Participants | 13 | 7
Statistical Analysis 1: Comparison: Experimental Treatment vs Active Comparator; Test type: Superiority; p = 0.35, t-test, 2 sided

6. Primary Outcome: Post-Study Usability Ratings
Description: An exit poll with 25 items was used to evaluate acceptability and usefulness ratings of the intervention:
  Sixteen items assessed Acceptability Rating of the WASABI app with a Likert scale from (1) Completely Disagree to (7) Completely Agree. The Acceptability Rating score is out of 7, higher number is better. The reported Acceptability Rating score is an average of all scores.
  Nine items explored the Usefulness of content delivered during the group tele-therapy sessions and through cognitive assessments and EMAs with a Likert scale from (1) Not at all to (4) Extremely). The Usability Rating score is out of 4, higher number is better. The reported Usefulness Rating score is an average of all scores.
Time Frame: At end of 16 weeks
Population: Data was only collected from the dCBGT+WASABI group (Experimental Treatment group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Treatment
Number analyzed (Participants) | 13
score on a scale
  Acceptability Rating Score | 5.1 (1.1)
  Usability Rating Score | 3.3 (0.6)

7. Primary Outcome: Reported Number of Adverse Effects
Description: The reported number of adverse events due to program use will be evaluated.
Time Frame: 16 weeks
Measure: Number; unit: adverse effects reported
Arm/Group | Experimental Treatment | Active Comparator
Number analyzed (Participants) | 13 | 7
adverse effects reported | 0 | 0
Statistical Analysis 1: Comparison: Experimental Treatment vs Active Comparator; Test type: Superiority; p = 0.95, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data are collected throughout the study duration. Study participation is 16 weeks.
Description: Adverse events are assessed at each assessment visit (at Baseline and Post-Intervention vists) and throughout the intervention period.
Arm/Group | Experimental Treatment | Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7

LIMITATIONS AND CAVEATS:
Lack of diversity in study population, 4 participants from ethnic groups withdrew prior to randomization. We did not record information on the time spent by the WASABI clinician in monitoring engagement, progress, and in providing feedback beyond the weekly group sessions. Since the WASABI group filled out 16 SPAI items many more times than the control group, this can could potentially limit the scientific rigor of the results. Using only one clinician as the therapist for all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03990870/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT03990870/SAP_001.pdf